CLINICAL TRIAL: NCT02698904
Title: A Quick Relaxation Training for People With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Relaxation Training for People With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDG_COPDRELAX_01
Record Dates: First submitted 2016-02-23; First posted 2016-03-04 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2016-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease (COPD); Relaxation Technique; Anxiety
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Anxiety Disorders | interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Guided Relaxation Technique (Experimental): Forced Vital Capacity (FVC), Forced Expiratory Volume in the First Second (FEV1), FEV1/FVC, Heart Rate Variability (HRV), airway resistance (kPa/l/s), before and after an 11 minutes, one-session, guided relaxation technique Following 30-40 minutes questionnaire, 5 minutes heart rate (HR) and oxygen saturation (SpO2) recording, 11 minutes relaxation technique (listening via headphone to audio recording. In the meanwhile, heart rate and saturation are recording) to be completed by second heart rate (HR) and oxygen saturation (SpO2) recording. Entire procedure 60-80 minutes.
  Interventions: Behavioral: Guided Relaxation Technique
- Documentary movie (Sham Comparator): Forced Vital Capacity (FVC), Forced Expiratory Volume in the First Second (FEV1), FEV1/FVC, Heart Rate Variability (HRV), airway resistance (kPa/l/s), before and after an 11 minutes documentary movie.
  Following 30-40 minutes questionnaire, 5 minutes heart rate (HR) and oxygen saturation (SpO2) recording, 11 minutes documentary movie (listening via headphone. In the meanwhile, heart rate and saturation are recording) to be completed by second heart rate (HR) and oxygen saturation (SpO2) recording. Entire procedure 60-80 minutes.
  Interventions: Other: Documentary Movie

INTERVENTIONS:
Behavioral: Guided Relaxation Technique
  Other Names: Relaxation Therapy
  Arms: Guided Relaxation Technique
Other: Documentary Movie
  Arms: Documentary movie

SUMMARY:
People with Chronic Obstructive Pulmonary Disease (COPD) suffer from dyspnoea, which may be exacerbated by psychological outcomes including anxiety and depression. Previous studies suggest that relaxation techniques may have positive effects on pulmonary rehabilitation. The main aim of this study is to explore both the respiratory and psychological impact of a quick, one-session, relaxation training for people with Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent;
* Chronic Obstructive Pulmonary Disease (COPD) diagnosis confirmed by a specialized physician;
* basal FEV1/FVC <70%, using the standards established by Global Initiative For Chronic Obstructive Lung Disease (GOLD);
* Modified British Medical Research Council Questionnaire (mMRC) ≥ 2;
* COPD Assessment Test (CAT) ≥ 10.

Exclusion Criteria:

* Pregnancy;
* psychiatric disturbances;
* oncological diseases;
* comorbid states that determine an immunosuppressive condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Differences in patients' state of dyspnea, before and after the treatment, as assessed by the Borg Scale (BORG) | Baseline and following filling in all the psychological tests and the session of relaxation technique/documentary movie (60-80 minutes elapsed time)

SECONDARY OUTCOMES:
Changes in Heart Rate Variability (HRV), before, during and after the treatment | It is recorded for 5 minutes before, during and after the session of relaxation technique/documentary movie (60-80 minutes elapsed time)
Changes in oxygen saturation (SpO2), before, during and after the treatment | It is recorded for 5 minutes before, during and after the session of relaxation technique/documentary movie (60-80 minutes elapsed time)
Changes in airway resistance (kPa/l/s) before and after the treatment | Baseline and following filling in all the psychological tests and the session of relaxation technique/documentary movie (60-80 minutes elapsed time)
Changes in subjective feelings of anxiety, before and after the treatment, as measured by the State Trait Anxiety Inventory (STAI-Y1) | Before the session of relaxation training/documentary movie and after it (60-80 minutes elapsed time)
Changes in the intensity of subjective feelings, before and after the treatment, as assessed by a Visual Analogue Scale (VAS) | Before the session of relaxation training/documentary movie and after it (60-80 minutes elapsed time)
Changes in the intensity of positive and negative affects, before and after the treatment, as assessed by the Positive and Negative Affective Schedule (PANAS) | Before the session of relaxation training/documentary movie and after it (60-80 minutes elapsed time)
Presence and intensity of the possible subjective experience of engaging just-manageable challenges by tackling a series of goals, continuously processing feedback about progress, and adjusting action based on this feedback, after the treatment | After the session of relaxation training/documentary movie (60-80 minutes after the baseline)
  Presence and intensity of the possible state of flow experience, as assessed by a short form of the Flow State Scale, called Short Flow State Scale -2 (FSS-2)
Differences in Forced Vital Capacity (FVC), before and after the treatment | Baseline and following filling in all the psychological tests and the session of relaxation technique/documentary movie (60-80 minutes elapsed time)
Differences in Forced Expiratory Volume in The First Second (FEV1), before and after the treatment | Baseline and following filling in all the psychological tests and the session of relaxation technique/documentary movie (60-80 minutes elapsed time)

CONTACTS AND LOCATIONS:
Locations (1):
- Paolo Banfi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Volpato E, Banfi P, Nicolini A, Pagnini F. A quick relaxation exercise for people with chronic obstructive pulmonary disease: explorative randomized controlled trial. Multidiscip Respir Med. 2018 May 2;13:13. doi: 10.1186/s40248-018-0124-9. eCollection 2018. PMID 29744054